CLINICAL TRIAL: NCT00713986
Title: Non-Pharmacologic Interventions to Relief Pain in Healthy Newborns Submitted to Vaccination to Hepatitis B: a Comparison Between Skin-to-Skin Contact, Glucose 25% and Both of Them
Brief Title: Non-Pharmacologic Interventions to Relief Pain in Healthy Newborns Submitted to Vaccination to Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Ruth Guinsburg, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID: AGC 1107
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2008-07-14 (Estimated); Status verified 2008-07

CONDITIONS: Pain; Analgesia
Keywords: Pain; Newborn Infant; Analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Water; Glucose; Lead; Tin Fluorides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Noanalgesia (Sham Comparator): Patients in this group wil receive 2 mL of water PO 2 minutes prior to vaccination, then they will rest in crib during cleansing of the right tigh, during injection of the right tigh for hepatitis B vaccination and 2 minutes after the injection. Infants will not receive any handling during the whole procedure outside the prespecified above.
  Interventions: Procedure: Water 2mL PO 2 minutes prior to intra-muscular injection
- Skin-to-skin (Experimental): Patients in this group wil receive 2mL of water 2 minutes prior vaccination and will be put on skin-to-skin contact with their mothers at the same time. After this time cleansing of the right tigh will be done followed by intra-muscular injection for hepatitis B vaccination. Patients will stay on skin-to-skin contact with their mothers for the following 2 minutes after injection. Infants will not receive any additional sensorial stimulation during the whole procedure outside the prespecified above.
  Interventions: Procedure: skin-to-skin contact
- Glucose (Experimental): Patients in this group wil receive 2mL of glucose 25% 2 minutes prior vaccination, then they will rest in crib during cleansing of the right tigh, during injection of the right tigh for hepatitis B vaccination and 2 minutes after the injection. Infants will not receive any handling during the whole procedure outside the prespecified above.
  Interventions: Procedure: Glucose 25% 2 mL PO 2 minutes prior to injection
- Skin&Glucose (Experimental): Patients in this group wil receive 2mL of glucose 25% PO 2 minutes prior vaccination and will be put on skin-to-skin contact with their mothers at the same time. After this time cleansing of the right tigh will be done followed by intra-muscular injection for hepatitis B vaccination. Patients will stay on skin-to-skin contact with their mothers for the following 2 minutes after injection. Infants will not receive any additional sensorial stimulation during the whole procedure outside the prespecified above.
  Interventions: Procedure: neonates will receive skin-to-skin contact beginning 2 minutes after the intra-muscular injection and stopping 2 minutes afterwards.

INTERVENTIONS:
Procedure: Water 2mL PO 2 minutes prior to intra-muscular injection — Sterile Water 2mL PO - single dose
  Arms: Noanalgesia
Procedure: skin-to-skin contact — neonates will receive skin-to-skin contact beginning 2 minutes before the intra-muscular injection and stopping 2 minutes afterwards.
  Arms: Skin-to-skin
Procedure: Glucose 25% 2 mL PO 2 minutes prior to injection — Glucose 25% 2mL PO - single dose
  Arms: Glucose
Procedure: neonates will receive skin-to-skin contact beginning 2 minutes after the intra-muscular injection and stopping 2 minutes afterwards. — neonates will receive 2 mL of glucose 25% PO (single dose) 2 minutes prior to the acute painful procedure. Skin-to-skin contact will start 2 minutes after the intra-muscular injection and will stop 2 minutes afterwards.
  Arms: Skin&Glucose

SUMMARY:
Acute procedural pain in neonates may be alleviated by non-pharmacological procedures. This study objective is to test the efficacy regarding pain attenuation of 3 interventions (skin-to-skin contact versus glucose 25% versus skin to skin associated to glucose 25) versus control in healthy newborn infants submitted to intra-muscular vaccination for Hepatitis B at 48-72 hours of life.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Gestational age of 37 0/7 to 41 6/7 weeks.
* Patients cared in rooming-in, with post-natal age of 12 to 72 hours of life.
* Adequate for gestational age and healthy infants.
* No other painful stimuli before study except for Vitamine K injection soon after birth.
* Interval from last feeding between 30 and 60 minutes.

Exclusion Criteria:

* Mothers that used opioid at gestation labor or birth.
* Delivery under general anesthesia.
* Apgar score less than seven in the 1st or 5th minute of life.
* Neonates that received any venous, arterial, capillary or spinal puncture.
* Any congenital malformation or CNS abnormality.

Ages: 12 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 640 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Neonatal pain scales: Neonatal infant pain Scale (NIPS), Neonatal Facial Coding System (NFCS) and Premature Infant Pain Profile (PIPP) | before the pain procedure (atrest), during cleaning of the region, at injection, and 2 minutes after injection

SECONDARY OUTCOMES:
Physiologic pain assessment variables: heart rate and oxygen saturation | before the pain procedure (atrest), during cleaning of the region, at injection, and 2 minutes after injection

CONTACTS AND LOCATIONS:
Overall Officials: Aurimery G Chermont, Principal Investigator — Federal University of Para and Federal University of São Paulo; Ruth Guinsburg, Study Director — Federal University of São Paulo

REFERENCES:
- [Derived] Chermont AG, Falcao LF, de Souza Silva EH, de Cassia Xavier Balda R, Guinsburg R. Skin-to-skin contact and/or oral 25% dextrose for procedural pain relief for term newborn infants. Pediatrics. 2009 Dec;124(6):e1101-7. doi: 10.1542/peds.2009-0993. PMID 19948613